CLINICAL TRIAL: NCT07035886
Title: Post-Marketing Surveillance (Usage Results Study) of Fruzaqla Capsule (Fruquintinib) for the Approved Indications in South Korea
Brief Title: A Study to Monitor the Fruzaqla Treatment of Adults With Metastatic Colorectal Cancer (mCRC) in South Korea
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-113-4001
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer
Keywords: Fruzaqla; Fruquintinib; Non-interventional
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- All Study Participants: Data will be collected for participants with metastatic colorectal cancer (mCRC) who will receive Fruzaqla according to the approved indication as per the Physician's routine schedule.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — As this is an observational study, no intervention will be administered.

SUMMARY:
The purpose of this study is to estimate the proportion of all adverse events (AEs) including serious adverse events (SAEs) occurring with the use of fruquintinib among adult participants who have been administered fruquintinib as per the approved indications.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to (>=)18 years.
* Participants who are initiate treatment or will be treated with Fruzaqla according to the approved label of South Korea.
* Participant voluntarily consent to participate in the study.

Exclusion criteria:

* Participants for whom Fruzaqla is contraindicated or those with risks that should avoid starting Fruzaqla, as per the product label.
* Participants actively participating in other interventional clinical trial(s) on mCRC treatments.
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with mCRC in South Korea who initiate the first treatment with Fruzaqla according to the approved indication will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Any Adverse Events (AEs), Adverse Drug Reaction (ADRs), Expected and Unexpected AEs and ADRs | Up to approximately 6 years
Number of Participants with Any Serious Adverse Events (SAEs), Serious Adverse Drug Reaction (SADRs), Expected and Unexpected SAEs and SADRs, AEs Leading to Death | Up to approximately 6 years
Number of Participants with AEs with Grade 3 or Higher | Up to approximately 6 years
Number of Participants who Reported the Events Related to Important Risks in the Risk Management Plan (RMP) | Up to approximately 6 years

SECONDARY OUTCOMES:
Overall Survival (OS) Rate | Up to 6 months
  OS rate is the percentage of participants who are alive for 6 months after their start date of Fruzaqla capsule.
Progression Free Survival (PFS) Rate | Up to 6 months
  PFS rate is the percentage of participants who have not experienced progression or death for 6 months after their start date of Fruzaqla capsule.
Objective Response Rate (ORR) | Up to 18 treatment cycles (approximately up to 18 months)
  ORR is defined as the percentage of participants achieving a best response of complete response (CR) or partial response (PR).
Disease Control Rate (DCR) | Up to 18 treatment cycles (approximately up to 18 months)
  DCR is defined as the percentage of participants achieving a best response of CR, PR, or Stable Disease (SD).
Median Overall Survival (mOS) | Up to 18 treatment cycles (approximately up to 18 months)
  OS will be defined as the time from the start date of Fruzaqla to the date of death from any cause. The mOS is the time at which 50% of participants are expected to have died from any cause.
Median Progression Free Survival (mPFS) | Up to 18 treatment cycles (approximately up to 18 months)
  PFS will be defined as the time from the start date of Fruzaqla capsule to the date of documented progression or death from any cause. Tumor assessment will be performed by routine clinical practice of the investigators. The mPFS is the time at which 50% of participants are expected to have experienced disease progression or died from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Yonsei University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click this link. — https://clinicaltrials.takeda.com/study-detail/2c248929b3e44ca6??page=1&idFilter=TAK-113-4001